CLINICAL TRIAL: NCT02513056
Title: Prospective Observational Study Evaluating the Use of MRI on CMS Beneficiaries With Non-Conditional Pacemakers and/or Implantable Cardioverter Defibrillators
Brief Title: Study Evaluating the Use of MRI on CMS Patients
Acronym: PM/ICD
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 821487
Record Dates: First submitted 2014-12-08; First posted 2015-07-31 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Pacemaker; Implantable Cardioverter Defibrillators
Keywords: non-conditional pacemakers; implantable cardioverter defibrillator

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: MRI — MRI

SUMMARY:
The overall objective of this protocol is to evaluate the safety and utility of diagnostic MRI in Center for Medicare and Medicaid Services (CMS) beneficiaries with pacemakers and Implantable Cardioverter Defibrillators (ICD) and clinical need for MRI.

DETAILED DESCRIPTION:
A referring physician will request an outpatient MRI in an implanted device patient through an order placed in the electronic ordering system, over the telephone to the MRI scheduling office, or by directly contacting a radiologist or MRI technologist. Upon receiving such a request, the referring physician will be sent a copy of the attached screening form, which is used for all implanted device patients. The form includes instructions for obtaining approval for the study and space for documenting ordering physician, study indication, and information about the patient's implanted device (if their device is not followed by a UPHS physician). For CMS beneficiaries, an addition to the form will discuss the clinical trial and ask the referring physician how the results of the MRI will change patient treatment or prognosis and what would be done were an MRI not available. The approval of an attending radiologist in the radiology section that will be interpreting the study (e.g. neuroradiology for brain MRI, cardiovascular imaging for cardiac MRI) is required.

Once the patient is deemed eligible and consented, the study staff will enter the patient into the registry as well as register them onto the trial through PennChart.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are at least 18 years of age
2. Patients have a medically/clinically indicated need for an MRI as an outpatient
3. Patients with a non-MRI conditional pacemaker and/or ICD implanted after the year 2000
4. Patients are CMS beneficiaries
5. Patients are willing and able to sign consent and HIPAA authorization or is authorized to sign consent for subject.

Exclusion Criteria:

1. Other contraindications to MRI
2. Pacemaker or ICD implanted prior to the year 2000
3. Patient is unwilling/unable to sign consent and HIPAA authorization
4. Leads and/or generator implanted within 6 weeks of the proposed MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pacemakers and/or implantable cardioverter defibrillators (ICD) referred for an outpatient Magnetic Resonance Imaging (MRI) procedure.
Sampling Method: Non-Probability Sample
Enrollment: 872 (Actual)
Dates: Start 2015-08-17 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Physician decision making | 4 years
  The primary measure of this study is physician decision making. Referring physicians will be asked about the effect of the MRI clinical management strategy, planning of treatments and interventions, as well as if/how the MRI results prevented other diagnostic studies or interventions, and other exposures (such as to ionizing radiation or iodinated contrast from CT scans). Analysis will be tabulation of how scan would change treatment or prognosis and what would be done if MR not available (based upon referring physician response on the screening form, physician and how the physicians believe that having the MRI will impact the treatment and quality of life by completing the QOL form.

SECONDARY OUTCOMES:
Adverse Events | 4 years
  Adverse events related to the MRI scan will be recorded and reviewed. AE's will be reviewed based on the criteria set forth in the protocol. AEs will be documented on an AE form and AE log and then entered into a redcap database.

OTHER OUTCOMES:
Patients will be asked how the MRI affected their quality of life, concerning | 4 years
  Patients will complete a Quality of Life form identifying how the MRI affected their quality of life, concerning both the MRI procedure itself and the fact that the MRI could be performed and diagnostic information about their conditions obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Schnall, MD, PhD, Study Chair — University of Pennsylvania; Harold Litt, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States